CLINICAL TRIAL: NCT00031915
Title: Phase II Trial of Gleevec (Formerly Known as STI571) in Patients With Soft Tissue and Bone Sarcomas: A Multi-Disciplinary Trial of the North American Sarcoma Study Group of the Connective Tissue Oncology Society
Brief Title: Imatinib Mesylate in Treating Patients With Advanced Soft Tissue Sarcoma or Bone Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000069239; NCI-02-C-0097; CCUM-2001-034; CPMC-IRB-14060; NCT00029094 (obsolete NCT alias)
Record Dates: First submitted 2002-03-08; First posted 2003-01-27 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2003-10

CONDITIONS: Childhood Malignant Fibrous Histiocytoma of Bone; Sarcoma
Keywords: metastatic osteosarcoma; recurrent childhood rhabdomyosarcoma; recurrent osteosarcoma; embryonal childhood rhabdomyosarcoma; alveolar childhood rhabdomyosarcoma; pleomorphic childhood rhabdomyosarcoma; metastatic childhood soft tissue sarcoma; recurrent childhood soft tissue sarcoma; childhood fibrosarcoma; childhood synovial sarcoma; childhood liposarcoma; childhood alveolar soft-part sarcoma; childhood neurofibrosarcoma; childhood angiosarcoma; childhood malignant fibrous histiocytoma of bone; previously treated childhood rhabdomyosarcoma; metastatic Ewing sarcoma/peripheral primitive neuroectodermal tumor; recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor; fibrosarcomatous osteosarcoma
MeSH Terms: conditions — Sarcoma; Osteosarcoma; Fibrosarcoma; Liposarcoma; Hemangiosarcoma; Neuroectodermal Tumors, Primitive, Peripheral | interventions — Imatinib Mesylate

INTERVENTIONS:
Drug: imatinib mesylate

SUMMARY:
RATIONALE: Imatinib mesylate may stop the growth of tumor cells by blocking the enzymes necessary for cancer cell growth.

PURPOSE: Phase II trial to study the effectiveness of imatinib mesylate in treating patients who have metastatic or unresectable locally advanced soft tissue sarcoma or bone sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of imatinib mesylate, as measured by response rate, in patients with metastatic or unresectable locally advanced soft tissue or bone sarcoma who have failed one or more prior treatment regimens.
* Determine the clinical and laboratory toxic effects of this drug in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to disease subtype.

Patients receive oral imatinib mesylate twice daily. Treatment continues for 1 year in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 60-120 patients (6-12 per stratum) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed metastatic or unresectable locally advanced (stage IV or recurrent) soft tissue or bone sarcoma

  * Eligible subtypes:

    * Ewing's family (e.g., primitive neuroectodermal tumor)
    * Osteosarcoma
    * Synovial sarcoma
    * Rhabdomyosarcoma (e.g., alveolar, embryonal, or pleomorphic)
    * Liposarcoma (all variants)
    * Malignant fibrous histiocytoma
    * Peripheral nerve sheath (e.g., malignant peripheral nerve sheath tumor, neurofibrosarcoma, or schwannoma)
    * Fibrosarcoma
    * Angiosarcoma (all variants)
  * Failed standard therapy with no available salvage regimens
* Unidimensionally measurable target lesions by x-ray, CT scan, MRI, PET, or physical examination

  * Must be outside prior irradiation fields or have documented disease progression at least 6 weeks after completion of prior radiotherapy

PATIENT CHARACTERISTICS:

Age:

* 10 and over

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 3 times upper limit of normal (ULN)
* ALT and AST less than 2.5 times ULN

Renal:

* Creatinine less than 1.5 times ULN

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for at least 1 week after study participation for female patients and for at least 3 months after study participation for male patients

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* No hormonal birth control

Radiotherapy:

* See Disease Characteristics
* At least 3 weeks since prior radiotherapy and recovered

Surgery:

* Not specified

Other:

* At least 28 days since any prior systemic therapy

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-06; Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee J. Helman, MD, Study Chair — National Cancer Institute (NCI)
Locations (10):
- United States (10):
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - University of Texas - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Result] Chugh R, Wathen JK, Maki RG, Benjamin RS, Patel SR, Meyers PA, Priebat DA, Reinke DK, Thomas DG, Keohan ML, Samuels BL, Baker LH. Phase II multicenter trial of imatinib in 10 histologic subtypes of sarcoma using a bayesian hierarchical statistical model. J Clin Oncol. 2009 Jul 1;27(19):3148-53. doi: 10.1200/JCO.2008.20.5054. Epub 2009 May 18. PMID 19451433